CLINICAL TRIAL: NCT05008926
Title: The NIPA Study: A Randomized Double-blind Control Clinical Trial Naloxegol Administration to Prevent Opioids Induced Gastrointestinal Motility Disturbance in Brain Injured PAtients
Brief Title: The NIPA Study Naloxegol Administration to Prevent Opioids Induced Gastrointestinal Motility Disturbance in Brain Injured PAtients
Acronym: NIPA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29BRC18.0262 (NIPA)
Record Dates: First submitted 2021-08-10; First posted 2021-08-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Brain Injuries
Keywords: Impaired gastrointestinal transit; Subarachnoid Hemorrhage; Traumatic brain injury
MeSH Terms: conditions — Brain Injuries; Subarachnoid Hemorrhage; Brain Injuries, Traumatic | interventions — naloxegol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naloxegol (Experimental): Administration of Naloxegol 25 mg per day by nasogastric tube (NG) or orogastric tube (OG). The administration should be started within the first 24 hours after the patient is admitted to intensive care unit and continued for the duration of the administration of the morphine derivative and until 48 hours after its discontinuation.
  Management of constipation and gastroparesis according to the recommendations.
  Interventions: Drug: Naloxegol
- Placebo (Placebo Comparator): Administration of the placebo according to the same procedures as the experimental arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naloxegol — Administration of Naloxegol 25 mg per day by nasogastric tube (SNG) or orogastric tube (SOG). The administration should be started within the first 24 hours after the patient is admitted to intensive care and continued for the duration of the administration of the morphine derivative and until 48 hours after its discontinuation.
  Arms: Naloxegol
Drug: Placebo — Administration of the placebo according to the same procedures as the experimental arm.
  Arms: Placebo

SUMMARY:
Impaired gastrointestinal transit (IGT) especially constipation, is common among patients under mechanical ventilation, occurring in up to 80 % of the patients during the first week, and has been associated with worse outcome in intensive care unit (ICU). Although IGT in critically ill patients is multifactorial and some components are due to complex disease, there is increasing evidence that exogenous opioids contribute to bowel dysmotility.

Sedatives and especially opioids are largely used in the brain injured population to control intracranial pression, reduce metabolic rate, manage or prevent seizures, and improve mechanical ventilator synchrony. Therefore, brain injured patients are particularly at risk to develop IGT. The occurrence of IGT is associated with adverse outcomes in intensive care unit. Both gastric reflux and impaired peristaltic contractions are associated with ventilator-acquired pneumonia.

The actual challenge is to prevent motility disorders before it occurs. A preventive strategy could in turn reduce the occurrence of complications related to impaired gastrointestinal transit such as ventilator-acquired pneumonia, bacteremia etc. It could also reduce the complications of feed intolerance and thus reduce morbidity and mortality in ICU.

Naloxegol is a polyethylene glycol derivative of naloxol, which is a derivative of naloxone and a peripherally acting µ-opioid receptor antagonist. Contrary to naloxone, naloxegol has a very low penetration into the central nervous system, therefore it could be a relevant option for ileus prevention without the risk of impaired sedation.

The aim of our study is to assess the efficacy of the administration of naloxegol on the onset of early constipation and early ventilator-acquired pneumonia in brain injured patients receiving opioids for analgosedation.

DETAILED DESCRIPTION:
Multicenter, randomized, double-blind, placebo-controlled experimental study of Naloxegol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ to 18 years old
2. Admission to intensive care unit for traumatic brain injury or subarachnoid hemorrhage without other life-threatening injury
3. Patients under sedation with administration of opiate-agonists, μ receptor agonists (Sufentanil, Fentanyl, Remifentanil, Morphine) for less than 24 hours
4. Expected duration of invasive mechanical ventilation and sedation of 48 hours or more
5. Intracranial pressure monitoring
6. Enteral feeding by oro / nasogastric tube
7. Affiliated or beneficiary of the French social security system

Exclusion Criteria:

1. Patient who received opioids for more than 24 hours
2. Patient with refractory intracranial hypertension at the time of inclusion: intracranial hypertension requiring therapy other than analgo-sedation (thiopental, targeted temperature management, decompressive craniectomy)
3. Acute or chronic renal failure with creatinine clearance <60ml / min
4. Known or suspected acute gastrointestinal obstruction
5. Risk of digestive perforation:

   * history of peptic ulcer
   * Crohn's disease
   * Ogilvie syndrome
   * acute diverticulitis
   * infiltrating gastrointestinal tumor
   * recurrent or advanced ovarian cancer
   * peritoneal metastasis
   * recent abdominal trauma with risk of digestive perforation
6. Concomitant treatment with a strong or moderate inhibitory effect of CYP 3A4 (For example: clarithromycin, ketaconazole, itraconazole, telithromycin, ritonavir, indinavir, saquinavir) or with a strong inducing effect (carbamazepin, rifampicin, millepertuis)
7. Concomitant treatment with vascular endothelial growth factor (VEGF) inhibitor
8. Allergy to Naloxegol or one of its excipients
9. Recent history of myocardial infarction within the past 6 months, symptomatic congestive cardiovascular disease, QT ≥ 500 msec
10. Patient with a medical decision for rapid palliative care
11. Pregnancy and / or breastfeeding
12. Child Pugh C stage cirrhosis
13. Patient under legal protection or deprived of liberty
14. Patient with another life-threatening injury
15. History of clinically important alterations of the blood-brain barrier: primary brain tumors, metastasis or other inflammatory pathologies in the CNS, active multiple sclerosis, Alzheimer's disease at an advanced stage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of bowel movement | 6 days
Incidence of ventilator-acquired pneumonia | 7 days

SECONDARY OUTCOMES:
Proportion of patient-days who received the daily calorie goal (25 Kcal / kg / day) | 10 days
Number of patients who required one or more administration of erythromycin and / or metoclopramide for vomiting occurring during enteral feeding | 10 days
Number of patients who received one or more rectal laxative for constipation | 10 days
Time in days of occurrence of the first bowel movement (in case of late constipation) | 10 days
Number of patients with ventilator-acquired pneumonia after D7 of invasive mechanical ventilationventilation (after D7 of invasive mechanical ventilation) | 10 days
Number of days without invasive mechanical ventilation | 10 days
Duration of hospitalization in intensive care unit | 10 days
Glasgow Outcome Scale Extended Score | 6 month
  The Glasgow Outcome Scale (GOS) is a comprehensive assessment scale for functional outcome that classifies a patient's condition into one of five categories: Death, Vegetative State, Severe Handicap, Moderate Handicap or Good Recovery. The extended GOS scale (GOSE) allows a more detailed classification into eight categories, thanks to a subdivision into two levels (lower and higher) of the categories "severe handicap", "moderate handicap" and "good recovery"
Number of patients who experienced an episode of intracranial hypertension requiring targeted temperature management, barbiturates, or decompression craniectomy. | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Huet, PU-PH, Principal Investigator — CHU Brest
Locations (11):
- France (11):
  - CHU de Bordeaux - Réanimation chirurgicale, Bordeaux, France
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU de Lille, Lille
  - CHU de Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Hôpital La Pitié Salpétrière (APHP), Paris
  - CHU de Strasbourg, Strasbourg
  - CHU Tours - Hôpital BRETONNEAU, Tours
  - CHU Tours - Hôpital TROUSSEAU, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement